CLINICAL TRIAL: NCT04580875
Title: Role of Minimally Invasive Surgery in Management of Penetrating Abdominal Trauma in Children
Acronym: MISinPAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: dr. Muhammad Abdelhafez Mahmoud, MD (Other)
Responsible Party: Sponsor-Investigator, dr. Muhammad Abdelhafez Mahmoud, MD, Lecturer of pediatric surgery, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: AlAzharMIS
Record Dates: First submitted 2020-09-29; First posted 2020-10-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2020-10

CONDITIONS: Penetrating Abdominal Trauma
Keywords: Children; Penetrating Abdominal Trauma; Laparoscopy; Minimally Invasive Surgery; Urgent Laparotomy; Negative Exploration
MeSH Terms: interventions — Minimally Invasive Surgical Procedures; Laparoscopy

STUDY DESIGN:
Intervention Model Description: Prospective cohort study. within the same facility, cases were enrolled consecutively but at some instances, in 2 or the 3 facilities at the same time, a portion of cases were managed simultaneously.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally invasive surgery (laparoscopy, laparoscopic-assisted procedures) (Active Comparator): This study will be conducted out at 3 pediatric surgery tertiary centers (Al-Azhar University hospitals in Cairo, Prince Mohammed bin Abdulaziz Hospital in Riyadh and Maternity & Children's Hospital in Bisha) on patients aged from 1-14 years presenting to the ER by stable penetrating abdominal trauma with significant clinical/radiologic findings, in the period from April 2017 to March 2022. Responders to initial resuscitation will be managed by minimally invasive surgery (laparoscopy and laparoscopic-assisted procedures). All patients enrolled in the study will give a written informed consent even for possible conversion to laparotomy if necessary.
  Interventions: Procedure: Minimally invasive surgery (laparoscopy and laparoscopic-assisted procedures) in both diagnosis and treatment of penetrating abdominal trauma in Children
- Conservative management (Active Comparator): patients aged from 1-14 years presenting to the ER by penetrating abdominal trauma with imsignificant findings will be managed conservatively.
  Interventions: Procedure: Minimally invasive surgery (laparoscopy and laparoscopic-assisted procedures) in both diagnosis and treatment of penetrating abdominal trauma in Children

INTERVENTIONS:
Procedure: Minimally invasive surgery (laparoscopy and laparoscopic-assisted procedures) in both diagnosis and treatment of penetrating abdominal trauma in Children

SUMMARY:
Exploratory laparotomy has been traditionally used for managing penetrating abdominal trauma (PAT). Currently, minimally invasive surgery (for diagnosis and treatment purposes) is a well-established and rapidly growing modality for dealing with penetrating abdominal trauma in stable children. Herein, we aimed to evaluate the effectiveness and outcomes and emphasize the importance of timely intervention by minimally invasive surgery for PAT possessing the potential to violate the peritoneum in stable pediatric victims.

This prospective study was carried out on 102 hemodynamically stable pediatric cases with highly suspicious penetrating abdominal trauma (caused by gunshot, stab, & accidental stab), admitted and managed by minimally invasive surgery (laparoscopy & laparoscopic-assisted procedures). Information recorded for analysis included demographic data, anatomical location of injury, organs affected, operative findings, operative time, need for conversion to laparoscopic-assisted approach, length of stay, complications, missed injury, and mortality rate.

A total of 102 pediatric cases with highly suspicious penetrating abdominal trauma (PAT) were managed by minimally invasive surgery (MIS). They were 62 males and 40 females with mean age of 7.3±0.6 years (range, 1-14 years). They included 39 cases of gunshot, 30 cases of stab abdomen, and 33 cases of accidental stab.

In this study, there was 100% accuracy in defining the injured organs with zero percent missed injuries in addition to effective therapeutic potential as regard the role of minimally invasive surgery in management of penetrating abdominal trauma in children.

Type of Study: Prospective cohort study

DETAILED DESCRIPTION:
Aim of the study:

Herein, the investigators aim to present our experience, evaluate the effectiveness & outcomes, and emphasize the importance of timely intervention by minimally invasive surgery in managing PAT highly suspicious to violate the peritoneum in hemodynamically stable children.

Review of literature:

* Different management modalities of penetrating abdominal trauma in children (conservative, routine exploratory laparotomy, Laparoscopy).
* Disadvantages of selective non-operative management (SNOM) and negative (non-therapeutic) laparotomy for penetrating abdominal trauma in children.
* Merits of diagnostic and therapeutic laparoscopy for penetrating abdominal trauma in children.

Patients and Methods:

This is a prospective study, will be conducted out at 3 pediatric surgery tertiary centers (Al-Azhar University hospitals in Cairo, Prince Mohammed bin Abdul-Aziz Hospital in Riyadh and Maternity & Children's Hospital in KSA) on pediatric patients presenting to the ER by penetrating abdominal trauma in the period from January 2015 to February 2021. Responders to initial resuscitation will be managed by minimally invasive surgery (laparoscopy and laparoscopic-assisted procedures). The total anatomical region of interest is defined as the cylindrical area bounded superiorly by the nipple line and the inferiorly by symphysis pubis. All patients enrolled in the study will give a written informed consent even for possible conversion to laparotomy if necessary. The study will be approved by the Institutional Review Board and ethics committee of the hospitals. All bullets and sharp objects will be removed during the procedures after optimum secure hemostasis. The main objective is to laparoscopically manage all PAT highly suspicious to violate the peritoneum.

Cases will be admitted, resuscitated, and stabilized as per pediatric advanced life support (PALS) and advanced trauma life support (ATLS) protocol guidelines, meanwhile, cases will be investigated by appropriate laboratory & radiologic studies. All patients will undergo E-FAST ultrasound and contrast abdominopelvic CT. Documented patients' data will include patient demographics, mechanism of injury, location of injury, pediatric trauma score (PTS) on admission (included weight, systolic blood pressure, mental status, airway condition, skeletal fracture, & open wounds), need for preoperative blood transfusion, surgical approach, operative findings, duration of hospital stay, complications, need for re-intervention, and follow-up period.

Institutes of the study:

A multicenter study at Pediatric Surgery Departments, Al-Azhar University hospitals in Cairo, Prince Mohammed bin Abdul-Aziz hospital (PMAH) in Riyadh, and Maternity & Children's hospital in KSA.

Number of cases: One-hundred-Two cases. Time frame: period of 5 years.

Ethical Consideration:

The protocol will be discussed and approved for clinical study by the Ethical Research Committee at PMAH and other participating hospitals. The procedures and the aim of the study will be clearly explained to the patient and the family. A written informed consent will be obtained before enrollment of the patients into the study. The family refusal to give consent for laparoscopic management is respected but does not deprive the patient from getting surgical care by exploration laparotomy.

Preoperative preparation:

All patients will be subjected to full clinical examination, rapid history taking, and necessary laboratory investigations (CBC, Coagulation profile, Liver and Renal Function tests, rapid serology for HBV, HCV, & HIV) and preoperative imaging (E-FAST, CT). They will be rapidly assessed and resuscitated. They will receive a dose of triple broad-spectrum antibiotics 30 min-1 hour before surgery.

Follow-up:

Patients were followed-up for median period of 52±17.12 months (range, 6-60 months) with no patients lost to follow-up. Ninety-two patients were reviewed at the office clinic and 10 patients were contacted by phone.

Statistical analysis:

Data were analyzed using the statistical package for social sciences (SPSS) version 24.0 (IBM Corp, IBM SPSS Statistics for Windows, Armonk, NY, USA). Continuous variables were expressed as mean± standard deviation (SD), range, and average while categorical variables were expressed as frequency count and percentage. Fisher's exact test was used for comparison of frequency counts/percentage. The t test was used for comparison of mean values. A two-sided p value less than 0.05 was considered statistically significant.

Discussion:

Discussion will focus on laparoscopic management of penetrating abdominal trauma in children. The results obtained from this study will be compared with each other and with that reported in the literature.

The discussion will focus on operative difficulties, operative time, conversion to directed laparotomy (laparoscopic-assisted procedure), and complications. It will compare results of this study with the results of others. Discussion will determine the most accurate management modality for penetrating abdominal trauma in children which offers the best outcome and least morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Children up to 14 years of age with penetrating trauma having the potential to violate the peritoneum,
* Hemodynamically stable, or
* Responded to initial resuscitation

Exclusion Criteria:

* Patients with blunt trauma,
* Penetrating trauma cases non-responding to initial resuscitation thus mandating urgent, laparotomy,
* Peritonitis,
* Sepsis,
* Patients older than 14 years,
* Cases requiring damage-control strategy.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Rate of missed injury (number & percent) | 1 week
  Rate of missed injury
Complications (number & percent) | 1 year
  Complications
Mortality rate (number & percent) | 3 years
  Mortality rate

SECONDARY OUTCOMES:
Operative time (in minutes) | 1 day (day of surgery)
  Operative time
Hospital stay (in days) | 2 weeks
  postoperative hospital stay
Follow-up period (in months) | 3 years
  Follow-up period

OTHER OUTCOMES:
Need for preoperative blood transfusion (number & percent) | 1 day (day of surgery)
  Need for preoperative blood transfusion

IPD SHARING:
Plan to Share IPD: Yes
Data are available for other researchers including methodology, figures, tables, results, and philosophy of discussion and the value this study add to the literature
Supporting Information: Study Protocol, SAP, ICF
Time Frame: August 2020 till indefinitely
Access Criteria: after the article became accepted and available online.